CLINICAL TRIAL: NCT01038882
Title: MIDAZOLAM EFFECTIVENESS TO THE SEDATION IN FLEXIBLE BRONCHOSCOPY. A RANDOMIZED STUDY
Brief Title: Randomized Study With Midazolam for Sedation in Flexible Bronchoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario La Fe (Other)
Responsible Party: ENRIQUE CASES VIEDMA, GENERALIDAD VALENCIANA. AGENCIA VALENCIANA DE SALUD
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: HLaFe 324/08
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Last update posted 2009-12-24 (Estimated); Status verified 2009-03

CONDITIONS: Sedation; Tolerance; Anxiety; Satisfaction
Keywords: sedation; midazolam; flexible bronchoscopy; tolerance
MeSH Terms: conditions — Anxiety Disorders; Personal Satisfaction | interventions — Midazolam

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Midazolam (Active Comparator): The patients of this arma receives midazolam before the flexible bronchoscopy to maintain conscious sedation
  Interventions: Drug: Midazolam
- Physiological serum (Placebo Comparator)
  Interventions: Other: Physiological serum

INTERVENTIONS:
Drug: Midazolam — Sedation started by injecting a 4 ml drug bolus with midazolam (0.07-0.1 mg/kg dose). Supplemental doses of midazolam (2 mg) were administrated at an interval of >2 min to maintain conscious sedation
  Arms: Midazolam
Other: Physiological serum — We started by injecting a 4 ml drug bolus and we ad supplemental doses (2 ml) to maintain the conscious sedation
  Arms: Physiological serum

SUMMARY:
The Flexible Bronchoscopy (FB) is a diagnostic and therapeutic procedure which is not usually tolerated by the patient. This makes the examination more difficult and a repetition of the examination, if necessary, resulting in a lower diagnostic performance.

Furthermore, there is nowadays little information with a highly obvious level about the relationship between sedation and the patient´s satisfaction with the FB.

Midazolam is one of the most commonly used sedatives at the beginning for its rapid onset property and brief duration of action with sedatives, anxiolytics and amnesia properties.

The principal aim of our study is to analyse if the use of a local anaesthetic with midazolam whilst performing an FB improves the quality of examination in terms of tolerance for the patient. It would also be of interest to know if there is an improvement in the acceptance of a second or further FB and if this improves the satisfaction of the Bronchoscopist as far as the examination performed is concerned.

DETAILED DESCRIPTION:
PATIENTS AND METHODS:

A randomized, prospective study has been carried out; double blind and controlled with placebo to be treated with midazolam. This included 152 patients, randomized into two groups: Group A - 79(51.9%) patients which received midazolam before the FB, and Group B - (49.1%) patients which received placebo. The patients were given a questionaire of 13 questions about different aspects of perception of the procedure after the respiratory endoscopy and another was given to the Bronchoscopist.

RESULTS:

Both groups started off with a similar assessment of fear and nervousness before the FB. Nevertheless, Group A gave a much higher score than Group B referring to variables related to symptoms and feeling. The patients´ cooperation was assessed by the Bronchoscopist in a similar way in both groups, although the length of the procedure and difficulty was higher in the group treated with placebo (Group B).

ELIGIBILITY:
Inclusion Criteria:

* Patients referred for diagnostic flexible bronchoscopy
* American Society of Anaesthesiology (ASA) class of risk I to III

Exclusion Criteria:

* Patients undergoing flexible bronchoscopy procedures such advanced techniques (autofluorescence, NBI, endobronchial ultrasound (EBUS)...)
* Psychological disorders
* Hypersensitivity to benzodiazepine
* Severe chronic obstructive pulmonary disease (FEV1 < 50% predicted value, requirement for oxygen therapy
* Unstable haemodynamic status (defined as a heart rate < 60 or > 120 and/or a systolic blood pressure < 100 or > 180 mmHG)
* Sings of systemic or pulmonary infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2008-10; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
To analyse if the use of a local anaesthetic with midazolam whilst performing an flexible bronchoscopy improves the quality of examination in terms of tolerance for the patient | February 2009

SECONDARY OUTCOMES:
To know if there is an improvement in the acceptance of a second or further flexible bronchoscopy and if this improves the satisfaction of the bronchoscopist as far as the examination performed is concerned | February 2009

CONTACTS AND LOCATIONS:
Overall Officials: ENRIQUE CASES-VIEDMA, MD, Principal Investigator — AGENCIA VALENCIANA DE SALUD
Locations (1):
- Hospital Universaitario La Fe, Valencia, Valencia, Spain

REFERENCES:
- [Result] González R, De-La-Rosa-Ramírez, Maldonado-Hernández A, Domínguez-Cherit G. Should patients undergoing a bronchoscopy be sedated? Acta Anaesthesiol Scand 2003; 47: 411-5. Pérez Negrin LM, Batista Martín JJ, Acosta Fernández O, Trujillo Castilla JL, Gonzalvo Hernández F. Subjetive tolerance to flexible bronchoscopy. Journal of Bronchology 2001; 8: 166-9. Ruiz López FJ, Valdivia Salas MM, Latour Pérez J, Ros Lucas LA, Fernández Suarez B, Sánchez Gascón F, Lorenzo Cruz M. Flexible bronchoscopy with only topical anesthesia. J Bronchol 2006; 13: 54-7. Stolz D, Prashant NC, Leuppi J, Pflimlin E, Tamm M. Nebulized lidocaine for flexible bronchoscopy: A randomized, double-blind, placebo-controlled trial. Chest 2005; 128: 1756-60. Honeybourne D, Babb J, Bowie P, Brewin A, Fraise A, Garrard C, Harvey J, Lewis R, Neumann C, Wathen CG, Williams T. British Thoracic Society guidelines on diagnostic flexible bronchoscopy. Thorax 2001; 56:(suppl I) i1-i21. Houghton CM, Raghuram A, Sullivan PJ, O´Driscoll R. Pre-medication for bronchoscopy: a randomised double blind trial comparing alfetanil with midazolam. Respir Med 2004; 98: 1102-7. Clark G, Licker M, Younossian AB, Soccal PM, Frey JG, Rochat T, Diaper J, Bridevaux PO, Tschopp JM. Titrated sedation with propofol or midazolam for flexible bronchoscopy: a randomised trial. Eur Respir J. 2009; 34: 1277-83. Stolz D, Kurer G, Meyer A, Chhajed PN, Pflimlin E, Strobel W, Tamm M. Propofol versus combined sedation in flexible bronchoscopy: a randomised non-inferiority trial. Eur Respir J. 2009; 34: 1024-30. Stolz D, Chhajed PN, Leuppi JD, Brutsche M, Pflimlin E, Tamm M. Cough suppression during flexible bronchoscopy using combined sedation with midazolam an hydrocodone: a randomised, double blind, placebo controlled trial. Thorax 2004; 59: 773-6. Chhajed PN, Wallner J, Stolz D, Baty F, Strobel W, Brutsche MH, Tamm M. Sedative drug requirements during flexible bronchoscopy. Respiration 2005; 72: 617-21.